CLINICAL TRIAL: NCT01173120
Title: Sub-study-A Phase IIIB Multicenter, Randomized, Double-Blind, Double-Dummy Study to Compare the Efficacy and Safety of Abatacept Administered Subcutaneously and Intravenously in Subjects With Rheumatoid Arthritis, Receiving Background Methotrexate, and Experiencing an Inadequate Response to Methotrexate
Brief Title: Methotrexate - Inadequate Response Device Sub-Study
Acronym: MTX-IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-174 (Sub study); 2007-005434-37 (EudraCT Number)
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abatacept Combination Product (ACP) (Experimental): Participants from the long-term period of study NCT00559585 who enrolled in the ACP substudy switched to administration of subcutaneous (SC) abatacept via the ACP for the duration of the substudy. Abatacept was administered SC using the ACP by the participant or caregiver on Substudy Day 1 and at weekly intervals thereafter. The ACP was a pre-filled liquid product device delivering 125 mg abatacept/device (125 mg/mL).
  Interventions: Device: Abatacept combination product (ACP)

INTERVENTIONS:
Device: Abatacept combination product (ACP) — Abatacept Solution, Subcutaneous, 125 mg/device, Weekly, 3 months
  Other Names: Orencia; BMS-188667

SUMMARY:
The purpose of this study is to determine the safety and acceptability of a device used in place of traditional syringes for abatacept self-injection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages ≥ 18
* Participants who are considered methotrexate inadequate responders (MTX-IR)
* 10 or more swollen joints (66 joint count) and 12 or more tender joints (68 joint count)
* Participants were to have been enrolled in the main MTX-IR study and been treated with open label abatacept for at least 3 months in the long term period

Exclusion Criteria:

* Participants who failed one or multiple anti-tumor necrosis factor (TNF) therapies
* Participants who meet diagnostic criteria for any other rheumatic disease (e.g., lupus erythematosus)
* Participants with active vasculitis of a major organ system (except for subcutaneous rheumatoid nodules)
* Participants with severe chronic or recurrent bacterial infections
* Participants who have received treatment with rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept Combination Product (ACP): Participants from the long-term period of the IM101-174 main study who enrolled in the ACP substudy switched to administration of subcutaneous (SC) abatacept via the ACP for the duration of the substudy. Abatacept was administered SC using the ACP by the participant or caregiver on Substudy Day 1 and at weekly intervals thereafter. The ACP was a prefilled liquid product device delivering 125 mg abatacept/device (125 mg/mL).
Period: Overall Study
Arm/Group | Abatacept Combination Product (ACP)
Started | 62
Switched Back to Main Study | 57
Discontinued ACP Substudy and Main Study | 5
Completed | 0
Not Completed | 62
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1
Not completed — Participant Decision | 2
Not completed — Switch-Administrative Reason By Sponsor | 33
Not completed — Switch-Participant Decision | 12
Not completed — Switch-Difficulty With Device | 12

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 51
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  North America | 62
Weight [Mean (Standard Deviation); unit: kg] | 86.3 (20.1)
Mean Duration of Disease [Mean (Standard Deviation); unit: years] | 7.4 (10.1)
Duration of Disease-Categorical [Number; unit: participants]
  ≤ 2 years | 28
  >2 - ≤5 years | 10
  >5 - 10 years | 7
  >10 years | 17
Number of Tender Joints [Mean (Standard Deviation); unit: tender joints] — Tender joints are an indicator of rheumatoid arthritis. The number of tender joints in a standard 68 joint count was evaluated. The number of tender joints ranges from 0 to 68, where an increased number of tender joints indicates increasing level of disease severity.
  tender joints | 31.6 (15.2)
Number of Swollen Joints [Mean (Standard Deviation); unit: swollen joints] — Swollen joints are an indicator of rheumatoid arthritis. The number of swollen joints in a standard 66 joint count was evaluated. The number of swollen joints ranges from 0 swollen joints to 66, where an increased number of swollen joints indicates increasing level of disease severity.
  swollen joints | 20.8 (8.2)
Participant Pain Assessment [Mean (Standard Deviation); unit: units on a scale] — The participant self-reported pain assessment is a core component of the American College of Rheumatology (ACR)scoring system, where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale, with 0 mm representing no pain and 100 mm representing the most pain possible.
  units on a scale | 64.2 (21.5)
Physical Function (Health Assessment Questionnaire Disability Index [HAQ-DI]) [Mean (Standard Deviation); unit: units on a scale] — The disability section of the full HAQ includes 20 questions that assess physical functions in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and other common activities. The questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. Higher scores=greater dysfunction. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered.
  units on a scale | 1.5 (0.7)
Participant Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Participant self-reported global rheumatoid arthritis assessment core component of the ACR scoring system, where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale, with 0 mm representing no pain and 100 mm representing the most pain possible.
  units on a scale | 61.6 (19.7)
Physician Global Assessment [Mean (Standard Deviation); unit: units on a scale] — Physician global rheumatoid arthritis assessment core component of the ACR scoring system, where increasing score indicates increasing level of severity as indicated on a 100 mm Visual Analog Scale, with 0 mm representing no pain and 100 mm representing the most pain possible.
  units on a scale | 62.0 (17.4)
High Sensitivity C-Reactive Protein (hs-CRP) Level [Mean (Standard Deviation); unit: mg/dL] — hs-CRP is an acute phase reactant protein that is a clinical marker for rheumatoid arthritis. Levels of hs-CRP can be used to determine the disease activity score.
  mg/dL | 1.7 (1.2)
Disease Activity Score (DAS 28) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a continuous disease measure that is a composite of 4 variables: the 28 tender joint count, the 28 swollen joint count, CRP levels, and participant assessment of disease activity measure on a visual analogue scale. The DAS28 has numeric thresholds that define high disease activity (>5.1), low disease activity (<3.2) and remission (<2.6). A clinically significant response=decrease in DAS28 score of >1.2 from baseline.
  units on a scale | 6.0 (0.8)
Rheumatoid Factor (RF) Status [Number; unit: participants] — RF is an autoantibody (antibody directed against an organism's own tissues) most relevant in rheumatoid arthritis. It is an antibody against the Fc portion of Immunoglobulin (Ig)G, which is itself an antibody. RF and IgG join to form immune complexes that contribute to the disease process. A positive value for RF was >20 IU/mL; a negative value for RF was ≤20 IU/mL.
  participants
    Positive | 46
    Negative | 16
Baseline Methotrexate Dose [Mean (Standard Deviation); unit: mg/wk] | 17.2 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Treatment-related SAEs, SAEs Leading to Discontinuation, Adverse Events (AEs), Treatment-related AEs, and AEs Leading to Discontinuation
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: ACP substudy Day 1 to last substudy assessment occurring prior to the 1st dose of non-ACP subcutaneous (SC) abatacept, assessed up to 12 months
Population: As-Treated Population, defined as all participants enrolled in ACP substudy who received at least 1 dose of SC abatacept administered via the ACP.
Measure: Number; unit: participants
Groups:
- Abatacept Combination Product (ACP): Participants from the long-term period of the IM101-174 main study who enrolled in the ACP substudy switched to administration of SC abatacept via the ACP for the duration of the substudy. Abatacept was administered using the ACP by the participant or caregiver on Substudy SC on Day 1 and at weekly intervals thereafter. The ACP was a prefilled liquid product device delivering 125 mg abatacept/device (125 mg/mL).
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
participants
  Deaths | 0
  SAEs | 2
  Treatment-related SAE | 0
  SAEs Leading to Discontinuation | 0
  AEs | 36
  Treatment-related AEs | 11
  AEs Leading to Discontinuation | 0

2. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Abatacept Over Time in the ACP Device Substudy
Description: Trough levels of abatacept were evaluated based upon serum samples. Day 1 pharmacokinetics were based on exposure to the pre-filled syringes and did not reflect abatacept exposure via the ACP device.
Time Frame: Days 1, 29, 57, 85, 169, and 253 of ACP substudy
Population: As-Treated Population, defined as all participants enrolled in ACP substudy who received at least 1 dose of SC abatacept administered via the ACP. Trough concentrations in participants who discontinued from the substudy were not summarized descriptively, but were included in the concentration listings.
Measure: Geometric Mean (Standard Deviation); unit: ug/mL
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
ug/mL
  Day 1 (prior to administration with ACP) (n =53) | 24.34 (15.56)
  Day 29 (n=52) | 27.61 (14.12)
  Day 57 (n=39) | 31.52 (14.49)
  Day 85 (n=47) | 27.46 (17.43)
  Day 169 (n=35) | 26.85 (14.55)
  Day 253 (n=5) | 24.41 (14.19)

3. Primary Outcome: Number of Participants With AEs of Special Interest in the ACP Device Substudy
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs including all infections, local injection reactions (prespecified), and systemic injection reactions (within 24 hours of dosing).
Time Frame: ACP substudy Day 1 to last substudy assessment occurring prior to 1st dose of non-ACP SC abatacept (administered once participants switched back to main study). For participants discontinuing both studies: Day 1 of ACP dosing to 56 days post last ACP dose
Population: As-Treated Population, defined as all participants enrolled in ACP substudy who received at least 1 dose of subcutaneous abatacept administered via the ACP.
Measure: Number; unit: participants
Groups:
- Abatacept Combination Product (ACP): Participants from the long-term period of the IM101-174 main study who enrolled in the ACP substudy switched to administration of subcutaneous abatacept via the ACP for the duration of the substudy. Abatacept was administered subcutaneously using the ACP by the participant or caregiver on Substudy Day 1 and at weekly intervals thereafter. The ACP was a pre-filled liquid product device delivering 125 mg abatacept/device (125 mg/mL).
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
participants
  Infections | 17
  Local injection reactions | 5
  Systemic injection reactions | 2

4. Primary Outcome: Number of Participants With Laboratory Test Results in Hematology Meeting the Criteria for Marked Abnormality in the ACP Device Substudy
Description: BL=baseline; LLN lower limit of normal; ULN=upper limit of normal. Marked abnormality criteria: Hemoglobin: >3 g/dL decrease from BL; Hematocrit: <0.75*BL; Erythrocytes: <0.75*BL; Platelets: <0.67*LLN/>1.5*ULN, or if BL <LLN, use 0.5*BL/<100,000 mm^3; Leukocytes: <0.75*LLN/ >1.25*ULN, or if BL<LLN, use <0.8*BL/>ULN, or if BL>ULN, use >1.2*BL/<LLN; neutrophils+bands: <1.0*10^3 c/uL; eosinophils: >0.750*10^3 c/uL; basophils: >400 mm^3; monocytes: >2000 mm^3; lymphocytes: <0.750*10^3 c/uL/ >7.50*10^3 c/uL.
Time Frame: ACP substudy Day 1 to last substudy assessment occurring prior to 1st dose of non-ACP SC abatacept (administered once participants switched back to main study). For participants discontinuing both studies: Day 1 of ACP dosing to 7 days post last ACP dose.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 50
participants
  Low hemoglobin (LLN=11.5 g/dL) | 1
  Low hematocrit (LLN=34%) | 1
  Low erythrocytes(LLN=3.8 x10*6c/uL) | 1
  Low platelets (LLN=140*10^9 c/L) | 0
  High platelets (ULN=450*10^9 c/L) | 0
  Low leukocytes (LLN= 3.8*10^3 c/uL) | 0
  High leukocytes (ULN = 10.6*10^3 c/uL) | 1
  Low neutrophils+bands(LLN=1.8*10^3 c/uL) | 0
  High eosinophils (ULN= 7*10^3 c/uL) | 0
  High basophils (ULN= 0.2*10^3 c/uL) | 0
  High monocytes (ULN=1*10^3 c/uL) | 0
  Low lymphocytes (LLN= 0.7*10^3 c/uL) | 3
  High lymphocytes(ULN=4.5*10^3 c/uL) | 0

5. Primary Outcome: Number of Participants With Liver Function Laboratories Meeting MA Criteria in the ACP Device Substudy
Description: Marked abnormality criteria: Alkaline phosphatase (ALP): >2* ULN, or if BL>ULN then use >3* BL; aspartate aminotransferase (AST): >3* ULN, or if BL>ULN then use >4* BL; alanine aminotransferase (ALT): >3* ULN, or if BL>ULN then use >4* BL; G-Glutamyl transferase (GGT): >2* ULN, or if BL>ULN then use >3* BL; Bilirubin: >2* ULN, or if BL>ULN then use >4* BL; blood urea nitrogen (BUN): >2* BL; creatinine: >1.5* BL
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 50
participants
  High ALP (ULN=400 U/L) | 0
  High AST (ULN=44 U/L) | 1
  High ALT (ULN=55 U/L) | 1
  High GGT (ULN=65 U/L) | 2
  High bilirubin (ULN=1.2 mg/dL) | 0
  High BUN (ULN=26 mg/dL) | 1
  High creatinine (ULN=1.5 mg/dL) | 1

6. Primary Outcome: Number of Participants With Electrolyte Laboratories Meeting MA Criteria in the ACP Device Substudy
Description: Marked abnormality criteria: Sodium (Na): <0.95*LLN/ >1.05*ULN, or if BL<LLN then use <0.95* BL or >ULN, or if BL>ULN then use>1.05* BL or <LLN; potassium (K): <0.9* LLN/>1.1*ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; (Cl): <0.9* LLN/>1.1* ULN, or if BL<LLN then use <0.9* BL or >ULN, or if BL>ULN then use>1.1* BL or <LLN; calcium (Ca): <0.8* LLN/>1.2* ULN, or if BL<LLN then use <0.75* BL or >ULN, or if BL>ULN then use>1.25* BL or <LLN; phosphorous (P): <0.75* LLN/ >1.25* ULN, or if BL<LLN then use 0.67* BL or >ULN, or if BL>ULN then use>1.33* BL or <LLN
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 50
participants
  Low Na (LLN=135 mEq/L) | 0
  High Na (ULN=148 mEq/L) | 0
  Low K (LLN=3.5 mEq/L) | 1
  High K (ULN=5.5 mEq/L) | 1
  Low Cl (LLN= 96 mEq/L) | 0
  High Cl (ULN=109 mEq/L) | 0
  Low Ca (LLN=8.4 mg/dL) | 0
  High Ca (ULN=10.6 mg/dL) | 0
  Low P (LLN=0.8 mg/dL) | 0
  High P (ULN 5.6 mg/dL) | 0

7. Primary Outcome: Number of Participants With Other Chemistry and Urinalysis Laboratories Meeting MA Criteria in the ACP Device Substudy
Description: MA criteria: serum glucose (Glu): <65 mg/dL/>220 mg/dL;fasting serum Glu: <0.8* LLN/>1.5*ULN,or if BL<LLN then use 0.8*BL or >ULN,or if BL>ULN then use >2.0*BL or <LLN;total protein: <0.9*LLN/>1.1*ULN,or if BL<LLN then use <0.9*BL or >UNL,or if BL>UNL then use >1.1*BL or <LLN; albumin: <0.9*LLN,or if BL<LLN then use <0.75 BL;uric acid: >1.5*ULN,or if BL>ULN then use >2*BL. Urinalysis (Urine protein,urine Glu,urine blood,leukocyte esterase,Red Blood Cells [RBCs], White Blood Cells [WBCs]):Use ≥2 when BL value missing or when pre-dose=0 or 0.5; use ≥3 when pre-dose=1, use ≥4 when pre-dose=2 or 3
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 50
participants
  Low Glu (n=50) | 2
  High Glu (n=50) | 2
  Low fasting Glu (LLN=65 mg/dL) (n=12) | 0
  High fasting Glu (ULN=115 mg/dL) (n=12) | 0
  Low protein (LLN=6 g/dL) (n=50) | 0
  High protein (ULN=8.5 g/dL) (n=50) | 0
  Low albumin (LLN=3.5 g/dL) (n=50) | 0
  High uric acid (ULN=8.7 mg/dL) (n=50) | 0
  High urine protein (normal=trace) (n=50) | 0
  High urine glucose (normal=negative) (n=50) | 2
  High urine blood (normal=negative) (n=50) | 2
  High leukocyte esterase (n=19) | 1
  High urine WBC (n=25) | 10
  High urine RBC (n=18) | 3

8. Primary Outcome: Mean Systolic Blood Pressure (SBP) Over Time in the ACP Device Substudy
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
mm Hg
  Day 1 before injection (n=62) | 128.1 (14.96)
  Day 85 (n=50) | 130.7 (17.08)
  Day 169 before injection (n=42) | 128.0 (13.61)
  Day 253 before injection (n=15) | 127.3 (16.63)
  Day 365 (n=4) | 135.3 (7.80)

9. Primary Outcome: Mean Diastolic Blood Pressure (DBP) Over Time in the ACP Device Substudy
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
mm Hg
  Day 1 before injection (n=62) | 76.4 (8.08)
  Day 85 (n=50) | 78.7 (9.99)
  Day 169 before injection (n=42) | 75.7 (9.31)
  Day 253 before injection (n=15) | 78.1 (8.29)
  Day 365 (n=4) | 77.5 (14.73)

10. Primary Outcome: Mean Heart Rate Over Time in the ACP Device Substudy
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
beats per minute
  Day 1 before injection (n=62) | 73.4 (10.18)
  Day 85 (n=50) | 74.0 (9.53)
  Day 169 before injection (n=42) | 73.4 (9.22)
  Day 253 before injection (n=15) | 76.9 (12.73)
  Day 365 (n=4) | 84.3 (4.79)

11. Primary Outcome: Mean Temperature Over Time in the ACP Device Substudy
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 62
degrees Celsius
  Day 1 before injection (n=62) | 36.6 (0.39)
  Day 85 (n=50) | 36.6 (0.36)
  Day 169 before injection (n=42) | 36.6 (0.39)
  Day 253 before injection (n=15) | 36.6 (0.27)
  Day 365 (n=4) | 36.4 (0.38)

12. Secondary Outcome: Number of Participants With Positive Anti-abatacept or Anti-Cytotoxic T Lymphocyte Antigen 4-T Cell (CTLA4-T) Responses Over Time by Enzyme Linked Immunosorbant Assay (ELISA) in the ACP Device Substudy
Description: Serum samples from all treated adult participants with active rheumatoid arthritis were screened for the presence of drug-specific antibodies using ELISA. Immunogenicity was defined as the presence of a positive anti-abatacept or anti-CTLA4 antibody.
Time Frame: ACP substudy Day 1 to last substudy assessment occurring prior to 1st dose of non-ACP SC abatacept (administered once participants switched back to main study). For participants discontinuing both studies: Day 1 of ACP dosing to 28 days post last ACP dose
Population: Immunogenicity Population, defined as all participants who received at least 1 dose of abatacept administered with the ACP who had at least one post Substudy Day 1 immunogenicity result available.
Measure: Number; unit: participants
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 53
participants
  Day 29 anti-ABA (n=50) | 0
  Day 29 anti-CTLA4 (n=51) | 0
  Day 29 total (n=51) | 0
  Day 57 anti-ABA (n=43) | 0
  Day 57 anti-CTLA4 (n=43) | 1
  Day 57 total (n=43) | 1
  Day 85 anti-ABA (n=42) | 0
  Day 85 anti-CTLA4 (n=42) | 0
  Day 85 total (n=42) | 0
  Overall on-treatment visits anti-ABA (n=53) | 0
  Overall on-treatment visits anti-CTLA4 (n=53) | 1
  Overall total on-treatment visits (n=53) | 1
  28 days post last dose anti-ABA (n=1) | 0
  28 days post last dose anti-CTLA4 (n=1) | 0
  28 days post last dose total (n=1) | 0
  Overall post visits anti-ABA (n=1) | 0
  Overall post visits anti-CTLA4 (n=1) | 0
  Overall post visits total (n=1) | 0
  Overall anti-ABA (n=53) | 0
  Overall anti-CTLA4 (n=53) | 1
  Overall total (n=53) | 1

13. Secondary Outcome: Number of Participants With Positive Anti-abatacept Responses Over Time by Electrochemiluminescence Immunoassay in the ACP Device Substudy
Description: An electrochemiluminescence immunoassay screened sera for drug-specific antibodies; immunocompetition was used to identify specific anti-Abatacept reactivity. CTLA4 and Possibly immunoglobulin (Ig) category=reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction (JNCT)category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity defined as a post-baseline titer higher than Baseline, or any post-baseline positivity if Baseline value was missing. TRT=treatment
Time Frame: ACP substudy Day 1 to last substudy assessment occurring prior to 1st dose of non-ACP SC abatacept (administered once participants switched back to main study). For participants discontinuing both studies: Day 1 of ACP dosing to 85 days post last ACP dose
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Abatacept Combination Product (ACP)
Number analyzed (Participants) | 60
participants
  Day 29 CTLA4 + possibly Ig (n=57) | 0
  Day 29 Ig and/or JNCT (n=57) | 1
  Day 29 total (n=57) | 1
  Day 57 CTLA4 + possibly Ig (n=47) | 0
  Day 57 Ig and/or JNCT (n=47) | 1
  Day 57 total (n=47) | 1
  Day 85 CTLA4 + possibly Ig (n=49) | 0
  Day 85 Ig and/or JNCT (n=49) | 0
  Day 85 total (n=49) | 0
  Day 169 CTLA4 + possibly Ig (n=43) | 0
  Day 169 Ig and/or JNCT (n=43) | 0
  Day 169 total (n=43) | 0
  Day 253 CTLA4 + possibly Ig (n=2) | 0
  Day 253 Ig and/or JNCT (n=2) | 0
  Day 253 total (n=2) | 0
  Overall on-TRT visits CTLA4 + possibly Ig (n=60) | 0
  Overall on-TRT visits Ig and/or JNCT (n=60) | 1
  Overall total on-TRT visits (n=60) | 1
  28 days post last dose CTLA4 + possibly Ig (n=1) | 0
  28 days post last dose Ig and/or JNCT (n=1) | 0
  28 days post last dose total (n=1) | 0
  56 days post last dose CTLA4 + possibly Ig (n=1) | 0
  56 days post last dose Ig and/or JNCT (n=1) | 0
  56 days post last dose total (n=1) | 0
  85 days post last dose CTLA4 + possibly Ig (n=1) | 0
  85 days post last dose Ig and/or JNCT (n=1) | 0
  85 days post last dose total (n=1) | 0
  Overall post visits CTLA4 + possibly Ig (n=1) | 0
  Overall post visits Ig and/or JNCT (n=1) | 0
  Overall post visits total (n=1) | 0
  Overall CTLA4 + possibly Ig (n=60) | 0
  Overall Ig and/or JNCT (n=60) | 1
  Overall total (n=60) | 1

ADVERSE EVENTS:
Arm/Group | Abatacept Combination Product (ACP)
Serious Adverse Events (participants affected / at risk) | 2/62
Other Adverse Events (participants affected / at risk) | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept Combination Product (ACP) (N=62)
Chest Pain (General disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept Combination Product (ACP) (N=62)
Bronchitis (Infections and infestations) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.